CLINICAL TRIAL: NCT01023178
Title: Comparison of Transdermal and Oral Estrogens in Adolescents With Ovarian Failure
Brief Title: Comparison of Transdermal and Oral Estrogens in Adolescent Girls With Ovarian Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Darrell M Wilson, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-10272009-4262
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Ovarian Failure, Premature
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Estradiol; Estrogens, Conjugated (USP); Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vivelle-Dot (Active Comparator): 17Beta Estradiol - transdermal
  Interventions: Drug: 17Beta Estradiol - transdermal; Drug: Progesterone, micronized
- Premarin (Active Comparator): Conjugated estrogens
  Interventions: Drug: Conjugated estrogens; Drug: Progesterone, micronized
- Estrace (Active Comparator): 17beta Estradiol
  Interventions: Drug: 17beta Estradiol; Drug: Progesterone, micronized

INTERVENTIONS:
Drug: 17beta Estradiol — Oral pill given daily at increasing doses every 6 months for 18 months.
  Other Names: Estrace
  Arms: Estrace
Drug: Conjugated estrogens — Oral pill, started at a low dose taken daily, dose increased every 6 months for 18 months
  Other Names: Premarin
  Arms: Premarin
Drug: 17Beta Estradiol - transdermal — Transdermal estrogen patch, started at low dose with increasing doses eery 6 months for 18 months
  Other Names: Vivelle-Dot
  Arms: Vivelle-Dot
Drug: Progesterone, micronized — Given starting at 18 months
  Other Names: Prometrium

SUMMARY:
To directly compare the safety (by laboratory evaluation) and efficacy (feminization and growth) of three commonly used estrogen preparations in adolescent patients with ovarian failure, either due to congenital causes (Turner syndrome) or medical therapies. We hypothesize that transdermal estrogen will have equivalent efficacy and a more favorable safety profile in comparison with conventional oral estrogen replacement.

DETAILED DESCRIPTION:
Treatment with transdermal 17beta(17β) estradiol resulted in higher estradiol levels and more effective feminization compared to oral conjugated equine estrogen but did not result in an otherwise different biochemical profile in this limited number of heterogeneous patients. OBE (oral beta estradiol) and TBE (transdermal beta estradiol) provide safe and effective alternatives to OCEE (oral conjugated equine estrogen) to induce puberty in girls, but larger prospective randomized trials are required.

ELIGIBILITY:
Inclusion Criteria: in whom initiation of estrogen therapy has been recommended due to ovarian failure

* Outpatients
* age >=12 years to 17.99 years old

Exclusion Criteria:

* spontaneous menses
* significant concurrent medical problem including:
* Liver function tests (LFTs) 3 times normal
* clotting disorder
* ongoing cancer treatment

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrell M Wilson, Principal Investigator — Stanford University; E Kirk Neely, Study Director — Stanford University; Sejal Shah, Sub-Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Shah S, Forghani N, Durham E, Neely EK. A randomized trial of transdermal and oral estrogen therapy in adolescent girls with hypogonadism. Int J Pediatr Endocrinol. 2014;2014(1):12. doi: 10.1186/1687-9856-2014-12. Epub 2014 Jun 20. PMID 24982681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from 2007-2011 study participants were recruited from pediatric endocrinology clinics at Lucile Packard Children's Hospital at Stanford.
Groups:
- Transdermal 17Beta Estradiol: 17Beta Estradiol - transdermal: Transdermal estrogen patch, started at low dose with increasing doses eery 6 months for 18 months
  Progesterone, micronized: Given starting at 18 months
- Oral Conjugated Equine Estrogen: Conjugated estrogens: Oral pill, started at a low dose taken daily, dose increased every 6 months for 18 months
  Progesterone, micronized: Given starting at 18 months
- Oral 17beta Estradiol: 17beta Estradiol: Oral pill given daily at increasing doses every 6 months for 18 months.
  Progesterone, micronized: Given starting at 18 months
Period: Overall Study
Arm/Group | Transdermal 17Beta Estradiol | Oral Conjugated Equine Estrogen | Oral 17beta Estradiol
Started | 5 | 8 | 7
Completed | 3 | 6 | 4
Not Completed | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal 17Beta Estradiol | Oral Conjugated Equine Estrogen | Oral 17beta Estradiol | Total
Number analyzed (Participants) | 5 | 8 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (0.5) | 13.8 (0.4) | 14.5 (0.6) | 14.2 (0.6)
Sex/Gender, Customized [Number; unit: participants]
  Female | 5 | 8 | 7 | 20
Follicle Stimulating Hormone (FSH) [Mean (Full Range); unit: mIU/mL] | 76 [1.5 to 144] | 86 [0.027 to 197] | 71 [0.656 to 144] | 78 [0.027 to 197]
Luteinizing Hormone (LH) [Mean (Full Range); unit: mIU/mL] | 14 [0.15 to 26] | 26 [0.009 to 86] | 13 [0.041 to 26] | 18 [0.009 to 86]

OUTCOME MEASURES:

1. Primary Outcome: Estradiol
Description: Estradiol blood levels at end of study compared across groups to determine effect of dosing methods. Significance of levels depends on the stage of puberty and goals of therapy.
Time Frame: end of study (up to 2 years)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Transdermal 17Beta Estradiol | Oral Conjugated Equine Estrogen | Oral 17beta Estradiol
Number analyzed (Participants) | 3 | 6 | 4
pg/mL | 53 (19) | 14 (5) | 12 (5)

ADVERSE EVENTS:
Arm/Group | Transdermal 17Beta Estradiol | Oral Conjugated Equine Estrogen | Oral 17beta Estradiol
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes